CLINICAL TRIAL: NCT03106233
Title: The Lateral Thigh Perforator (LTP) Flap for Autologous Breast Reconstruction: A Prospective Analysis of 138 Flaps
Brief Title: Lateral Thigh Perforator (LTP) Flap for Autologous Breast Reconstruction
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Rene van der Hulst, Prof. dr., Maastricht University Medical Center
Other Study IDs: METC 14-5-095
Record Dates: First submitted 2017-02-09; First posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer
Keywords: Breast reconstruction; Perforator flap; Microsurgery
MeSH Terms: conditions — Breast Neoplasms | interventions — Surgical Flaps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LTP flap breast reconstruction: All consecutive patients who underwent LTP flap breast reconstructions (unilateral, bilateral or stacked unilateral) between September 2012 and November 2016 at three centers in Maastricht, the Netherlands, and New York and New Orleans, the United States, were included. Autologous breast reconstruction was performed by using the upper lateral thigh region as a donor site.
  Interventions: Procedure: LTP flap

INTERVENTIONS:
Procedure: LTP flap — A flap is harvested from the upper lateral thigh region based on septocutaneous perforators located in the posterior septum between the tensor fascia latae and gluteus medius muscles.
  Other Names: Lateral thigh perforator flap; Septocutaneous tensor fasciae latae (sc-TFL) flap

SUMMARY:
The lateral thigh perforator (LTP) flap was previously introduced as an alternative flap for autologous breast reconstruction when the abdomen is not suitable as a donor site. In this prospective study all LTP flap breast reconstructions that have been performed since September 2012 are analyzed. In addition, the surgical refinements that were introduced over the years are reported.

ELIGIBILITY:
Inclusion Criteria:

* Lateral thigh region suitable as a donor site
* Abdomen not suitable as donor site
* Informed consent

Exclusion Criteria:

* Pre-operative imaging showing no suitable perforators

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only female participants
Study Population: All female patients who opted for autologous breast reconstruction but who required an alternate flap than the deep inferior epigastric artery perforator (DIEP) flap.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Recipient- and donor-site complications | Through study completion up to an average of 12 months post-operatively
  Recipient site: Total flap loss, partial flap loss, venous congestion, infection, hematoma, seroma, fat necrosis and wound complications. Donor site: Infection, hematoma, seroma, fat necrosis, wound complications.

SECONDARY OUTCOMES:
Flap re-explorations | Through study completion up to an average of 12 months post-operatively
  Total number of flaps that required a re-exploration because of arterial or venous insufficiency, hematoma or kinking of the pedicle.

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Tuinder, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided